CLINICAL TRIAL: NCT00153127
Title: Comparison of Braintree PolyethyleneGlycol(PEG) Laxative and Placebo for Relief of Constipation From Constipating Medications
Brief Title: Comparison of PolyethyleneGlycol and Placebo for Relief of Constipation From Constipating Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 851-17
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

INTERVENTIONS:
Drug: polyethyleneglycol3350

SUMMARY:
The purpose of this study is to assess treatment responses comparing a newly FDA-approved PEG laxative versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female ambulatory outpatient age 19 or older.
* Patients meet ROME II Criteria
* Patients not meeting ROME IBS criteria
* Use of a constipating medication (>= 3% in PDR)
* If female and of childbearing potential, patient must be surgically sterilized or using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study
* Written informed consent.

Exclusion Criteria:

* Known or suspected obstruction, gastric retention, ileus, perforation, fecal impaction or inflammatory bowel disease.
* Prior small bowel or colonic resection or colostomy.
* Weight < 80 lbs.
* Unwilling or unable to undergo any colon diagnostic examinations at the end of the study if not performed within 5 years of the informed consent date advised by clinically accepted indications.
* Positive stool hemoccult.
* Significant cardiac, renal or hepatic insufficiency.
* Pregnant or expecting to become pregnant within 120 days of study enrollment.
* Lactating or breast feeding.
* Subjects who in the opinion of the investigator would be unable to comply adequately with the study plan.
* Use of investigational drugs in the last 30 days.
* Patients with known allergy to PEG or PEG medications such as PEG or sulfate-free electrolyte lavage solutions

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-11; Primary Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
A successful outcome is defined as no longer meeting the definition of constipation using ROME I criteria

SECONDARY OUTCOMES:
Analysis of individual ROME I criteria
Safety (adverse event and laboratory testing)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Herrera, MD, Principal Investigator — University of South Alabama
Locations (4):
- United States (4):
  - Mobile, Alabama
  - St. Petersburg, Florida
  - St Louis, Missouri
  - Raleigh, North Carolina